CLINICAL TRIAL: NCT04753957
Title: Pharmacokinetics of Progesterone in Pregnancy-2
Acronym: PiP-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with endometrial sample collection. New study design to be prospective observational to validate reliable methods of endometrial sampling at time of c-section.
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20D.1094
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal progesterone (Active Comparator): 200mg micronized vaginal progesterone placed 7am prior to scheduled cesarean delivery
  Interventions: Drug: micronized Progesterone
- Control (No Intervention): No intervention, scheduled cesarean delivery

INTERVENTIONS:
Drug: micronized Progesterone — 200mg micronized progesterone placed vaginally
  Arms: Vaginal progesterone

SUMMARY:
The objective of this study is to evaluate the local pharmacokinetics of progesterone in pregnancy through evaluation of progesterone levels in maternal serum, endometrium, and cordblood in pregnant patients undergoing scheduled cesarean delivery.

DETAILED DESCRIPTION:
The objective of this pilot study is to evaluate the local pharmacokinetics of progesterone in pregnancy through evaluation of progesterone levels in maternal serum, endometrium, and cordblood in pregnant patients undergoing scheduled cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18yo
* Singleton gestation, ≥36 0/7 weeks gestation
* Scheduled cesarean delivery at Thomas Jefferson University Hospital or affiliate

Exclusion Criteria:

* Contraindication to vaginal progesterone suppository

  * Active hepatic disease
  * Prior or current thrombus
  * Known adverse reaction to progesterone
  * Peanut allergy
* Bleeding disorder (such as thrombophilia)
* Use of 17-hydroxyprogesterone caproate in the pregnancy
* Use of vaginal progesterone in the pregnancy
* History of adverse reaction to progesterone
* Current vaginitis

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Endometrial (ng/mg) progesterone time/concentration profile | 12 hours
  Concentration of progesterone in endometrium, sampled at time of scheduled c-section
Plasma (ng/ml) progesterone time/concentration profile | 12 hours
  concentration of serum progesterone, sampled at time of scheduled c-section

SECONDARY OUTCOMES:
Side effect survey | 24hr after delivery
  survey of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD may be requested following trial completion and publication with appropriate data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following trial completion and publication
Access Criteria: Data sharing agreement